CLINICAL TRIAL: NCT05897190
Title: Evaluate the Safety and Immunogenicity of a SARS-CoV-2 mRNA Vaccine (RBMRNA-405) as a Booster in Chinese Adults & Older
Brief Title: Evaluate the Safety and Immunogenicity of a SARS-CoV-2 mRNA Vaccine Booster
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Argorna Pharmaceuticals Co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CP-RBMRNA-001-01-P
Record Dates: First submitted 2023-05-28; First posted 2023-06-09 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: SARS-CoV-2
MeSH Terms: interventions — CVnCoV COVID-19 vaccine; sinovac COVID-19 vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SARS-CoV-2 mRNA vaccine (RBMRNA-405) adult group (Experimental): One dose was administered by intramuscular injection on day 1
  Interventions: Biological: SARS-CoV-2 mRNA vaccine (RBMRNA-405)
- SARS-CoV-2 mRNA vaccine (RBMRNA-405) older adult group (Experimental): One dose was administered by intramuscular injection on day 1
  Interventions: Biological: SARS-CoV-2 mRNA vaccine (RBMRNA-405)
- CoronaVac® adult group (Active Comparator): One dose was administered by intramuscular injection on day 1
  Interventions: Biological: CoronaVac®
- CoronaVac® older adult group (Active Comparator): One dose was administered by intramuscular injection on day 1
  Interventions: Biological: CoronaVac®

INTERVENTIONS:
Biological: SARS-CoV-2 mRNA vaccine (RBMRNA-405) — Dose A
  Arms: SARS-CoV-2 mRNA vaccine (RBMRNA-405) adult group; SARS-CoV-2 mRNA vaccine (RBMRNA-405) older adult group
Biological: CoronaVac® — Dose B
  Arms: CoronaVac® adult group; CoronaVac® older adult group

SUMMARY:
This study is to evaluate the safety and immunogenicity of a SARS-CoV-2 mRNA Vaccine as a heterologous booster dose in adults who completed 2 doses of inactivated vaccination through 12 months in China.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 years and older, Body Mass Index (BMI) is between 18-30, able to provide legal proof of identity
2. Participants voluntarily agreed to participate in the study and signed an informed consent form
3. The subject has the ability to understand the study process and is willing and able to comply with all study proposals and other requirements of the study
4. Be willing and able to comply with protocol and complete 12-month study follow-up
5. Have received 2 doses of inactivated SARS-CoV-2 vaccine for 6 months and less than 12 months before enrollment
6. Male and female subjects of childbearing age agree to use effective contraception from screening period until 12 months after vaccination; female subjects of childbearing age have taken effective contraceptive measures 1 month before enrollment
7. Female subjects of childbearing age are not at pregnant period (negative result of pregnancy test) or lactation period
8. Male and female subjects of child-bearing age agree that do not donate eggs (eggs, oocytes) for assisted reproduction (female subjects of reproductive age) or avoid sperm donation (male subjects) from screening period until 12 months after vaccination

Exclusion Criteria:

1. Have received any SARS-CoV-2 vaccines other than 2 doses of the inactivated vaccine
2. History of Severe Acute Respiratory Syndrome (SARS), Coronavirus disease 2019 (COVID-19), Middle East Respiratory Syndrome (MERS) and other human coronavirus infections or disease
3. Positive SARS-CoV-2 reverse transcription-polymerase chain reaction (RT-PCR) test
4. The vital signs or physical examination are clinically significant abnormal as determined by the investigators in screening
5. Fever (axillary temperature≥37.3°C) on the day of the vaccination
6. A history of severe allergy (including drugs, vaccines, and foods) or to any component of the experimental vaccine, e.g., allergic shock, laryngeal edema, anaphylactoid purpura, dyspnea, and angioedema, etc.
7. Subjects have contraindications to intramuscular injection, such as having been diagnosed with thrombocytopenia, any blood clotting disorder, or receiving anticoagulant therapy
8. Subjects have been diagnosed with a serious disease, congenital malformation or chronic disease (including but not limited to respiratory disease or bronchitis such as asthma, serious cardiovascular disease, serious cerebrovascular disease, kidney disease, serious or uncontrollable diabetes, autoimmune disease, thrombocytopenic purpura, thalassemia, malignant tumor, hereditary allergic constitution, etc.) that may interfere with the conduct or completion of the study
9. Diagnosed with diseases may affect immune system function, including malignant tumor, congenital or acquired immune deficiency or suppression (e.g., tuberculosis, human immunodeficiency virus (HIV)), Hepatitis B, hepatitis C, syphilis infection, uncontrollable autoimmune disease, no spleen or spleen dysfunction
10. History or family history of central nervous system disease, convulsions or tics, epilepsy, meningitis, neurological disorders, mental disorders, cerebritis, myelitis, Guillain-Barre syndrome, etc
11. Long-term use of immunopotentiator or immunosuppressant therapy within 6 months prior to vaccination (continuous oral or injection for more than 14 days)
12. Use of any blood or blood-related products (e.g., blood transfusion, use of human albumin, human immunoglobulin, etc.) or have received solid organ or bone marrow transplantation within 3 months prior to vaccination
13. Lymph node - related diseases (such as lymphadenitis, lymph node adhesion, lymph node tuberculosis, tumor metastasis, etc.) or skin scars and fistulas at the lymph node site, or lymphadenopathy, tenderness, skin redness and swelling at the lymph node site within 7 days prior to vaccination
14. Within 3 days prior to vaccination, an acute illness or attack of a chronic disease, or the use of antipyretic analgesic or anti - allergic drugs
15. Other vaccines have been administered within 4 weeks prior to the trial vaccination or other vaccination schedule (except for emergency vaccinations such as Rabies vaccine and Tetanus vaccine) between the screening period and 28 days after the vaccination
16. Participating in or planning to participate in other clinical trials (drugs or vaccines) within 3 months prior to participating in this study
17. Any blood loss >400 mL (e.g., donation of blood or blood components or injury) within 28 days prior to the screening visit, or plans to donate blood or blood components between the screening visit and 28 days post-vaccination
18. Any abnormal or permanent body art (such as tattoos) at the site of the vaccination, which the researchers think to interfere with observing local reactions at the site of the vaccination
19. Other circumstances considered by the investigator as inappropriate to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-05-16 (Actual); Primary Completion 2022-06-13 (Actual); Study Completion 2023-05-12 (Actual)

PRIMARY OUTCOMES:
Incidence of solicited local and systemic adverse events (AE) | Within 14 days after booster vaccination

SECONDARY OUTCOMES:
Incidence of serious adverse events (SAEs) | Within 360 days after booster vaccination
The levels of neutralizing antibodies anti-SARS-CoV-2 | The 14th day, 28th day after booster vaccination
The levels of Immunoglobulin G (IgG) antibody against the S protein of SARS-CoV-2 | The 7th day, 14th day, 28th day, 90th day, 180th day and 360th day after booster vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- Chengdu Xinhua Hospital affiliated to North Sichuan Medical College, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No